CLINICAL TRIAL: NCT03074760
Title: A Study of Acequias Contamination & Association of Infectious Diseases in Peru
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: BioRed LLC (Other)
Responsible Party: Sponsor
Other Study IDs: CUIRBRG273
Record Dates: First submitted 2017-03-04; First posted 2017-03-09 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Water-Related Diseases
MeSH Terms: conditions — Waterborne Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Contaminated acequias
  Interventions: Diagnostic Test: Adenovirus; Diagnostic Test: Rotavirus; Diagnostic Test: H. pylori
- Non-contaminated acequias
  Interventions: Diagnostic Test: Adenovirus; Diagnostic Test: Rotavirus; Diagnostic Test: H. pylori

INTERVENTIONS:
Diagnostic Test: Adenovirus — Diagnostic test for the presence of the adenovirus in the population groups
Diagnostic Test: Rotavirus — Diagnostic test for the presence of the Rotavirus in the population groups
Diagnostic Test: H. pylori — Diagnostic test for the presence of H. pylori infection in the population groups

SUMMARY:
A major water supply utilized in the Lambayeque region are acequias. Acequias are irrigation canals that are utilized by the agriculture industry for the cultivation of consumables. Utilization of contaminated water to irrigate consumables can lead to foodborne illnesses. Contamination studies on the acequias in the Lambayeque region have not been performed to date. The purpose of this study is to test contamination of acequias in 9 districts in Lambayeque and determine if a difference in infection rates exists in districts with contaminated acequias vs. districts without contaminated acequias for the following diseases: H. pylori, Adenovirus, Rotavirus.

ELIGIBILITY:
Inclusion Criteria:

* Currently reside in one of the following districts: Eten, Pomalca, Pimentel, Patapo, Pucala, Santa Rosa, Reque, Monsefu and Sana
* 18 years of age or older
* Consent to participate

Exclusion Criteria:

* Currently taking antiviral or antimicrobial medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There is no study population in phase I as it is focused on the districts and their corresponding acequias. Phase II of this study will include participants 18 years of age or older who consent to participate and are from the following districts: Eten, Pomalca, Pimentel, Patapo, Pucala, Santa Rosa, Reque, Monsefu and Sana.
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2017-03-16 (Actual); Primary Completion 2017-05-01 (Estimated); Study Completion 2017-05-01 (Estimated)

PRIMARY OUTCOMES:
Contamination of acequias | March 20th - April 1st
  Presence of Fecal Coliforms in the acequias

SECONDARY OUTCOMES:
Proportion of population with infections | March 20th - May 1st
  Proportion of populations with adenovirus, rotavirus and H. pylori infections

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Goode, Principal Investigator — Campbell University
Locations (5):
- Peru (5):
  - BioRed, Hacienda Pucala, Lambayeque
  - BioRed, Pátapo, Lambayeque
  - BioRed, Pimentel, Lambayeque
  - BioRed, Pomalca, Lambayeque
  - BioRed, Tumán, Lambayeque

IPD SHARING:
Plan to Share IPD: Undecided